CLINICAL TRIAL: NCT03486093
Title: Randomized Clinical Trial on the Role of Port Protectors for the Management of Venous Central Line Catheter in Respiratory Semi-intensive Care Unit.
Brief Title: Port Protectors for Prevention of CLABSIs in Respiratory Semi-intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Riccardo Inchingolo, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5664/13
Record Dates: First submitted 2018-03-07; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: Venous central catheter; Central line-associated bloodstream infections; Port protector; Respiratory semi-Intensive Care Unit

STUDY DESIGN:
Intervention Model Description: Patients have been randomized into two groups:
  1. patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations.
  2. Patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations with the aid of port protector devices.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVC managed by healthcare workers (Experimental): Patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations.
  Interventions: Behavioral: Training and retraining to GAVECELT "bundle" recommendations
- CVC managed by healthcare workers plus port protector (Experimental): Patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations with the aid of port protector devices.
  Interventions: Device: Training and retraining to GAVECELT "bundle" recommendations plus port protector

INTERVENTIONS:
Device: Training and retraining to GAVECELT "bundle" recommendations plus port protector — Physicians and nurses of RICU have been trained and retrained to GAVECELT "bundle" recommendations concerning the management of CVC. The bundle includes: hand hygiene and precautions for protection and safety, adequate insertion site, echo-guided placement of central venous line, use of clorexidine 2% for skin disinfection of insertion site chosen and subsequent continuous or discontinuous disinfection of exit site, use of suture-less devices, use of transparent semi-permeable dressing whenever applicable and immediate removal of catheter when no longer needed.
  After the first training meeting, the use of Curos® Disinfecting Port Protector for needleless valves port-protector has been introduced.
  Other Names: Curos® Disinfecting Port Protector for needleless valves port-protector (CUROS, 70% isopropyl alcohol-impregnated, Ivera Medical, San Diego, California, US).
  Arms: CVC managed by healthcare workers plus port protector
Behavioral: Training and retraining to GAVECELT "bundle" recommendations — Physicians and nurses of RICU have been trained and retrained to GAVECELT "bundle" recommendations concerning the management of CVC. The bundle includes: hand hygiene and precautions for protection and safety, adequate insertion site, echo-guided placement of central venous line, use of clorexidine 2% for skin disinfection of insertion site chosen and subsequent continuous or discontinuous disinfection of exit site, use of suture-less devices, use of transparent semi-permeable dressing whenever applicable and immediate removal of catheter when no longer needed.
  Arms: CVC managed by healthcare workers

SUMMARY:
Central Line-Associated BloodStream Infections (CLABSIs) are responsible for many deaths in the United States annually.

Several collaboratives have demonstrated the preventability of these infections.

Educational interventions decrease rates of CLABSIs. In addition to training, education, and surveillance, important prevention practices include the use of chlorhexidine skin antiseptics and maximal sterile barrier precautions at catheter insertion. Other maintenance practices include hand hygiene before handling catheters or catheter sites, chlorhexidine for skin antisepsis with dressing changes, and disinfecting catheter hubs or injection ports with an appropriate agent before accessing the catheter.

Antimicrobial catheter locks, including nonantibiotic antiseptic locks (such as alcohol or trisodium citrate), have also demonstrated some success in reducing CLABSIs. In particular, alcohol-impregnated port protectors and needleless neutral pressure connectors significantly reduced rates of CLABSIs.

Respiratory semi-intensive care units (RICUs) usually work as "step-up" units within acute care hospitals to manage patients with respiratory failure with non-invasive ventilation. These units may provide multidisciplinary rehabilitation and serve as a bridge to home-care programs or long-term care facilities. Some of these RICUs may work also as "step down" units for difficult to wean patients.

The investigators performed a single-centre prospective randomized clinical trial with the aim to assess the efficacy of educational interventions alone and combined with port protector as adjuvant tool on rate of CLABSIs. Moreover, the investigators evaluated the effects of previously mentioned interventions on rates of CVC colonizations and contaminated blood cultures.

DETAILED DESCRIPTION:
The study enrolled patients admitted to RICU and it lasted 18 months. Patients were enrolled when a CVC: 1) was placed during hospitalization in RICU; 2) had already been placed at admittance and patients didn't show signs of systemic inflammatory response syndrome (SIRS) during first 48h from admission to RICU; 3) had already been placed at admittance without evidence of microbiologic contamination of blood cultures.

Each patient gave written informed consent. Patients enrolled underwent blood cultures sampling whenever they showed SIRS signs.

SIRS is defined as 2 or more of the following variables: 1) fever of more than 38°C (100.4°F) or less than 36°C (96.8°F), 2) heart rate of more than 90 beats per minute, 3) respiratory rate of more than 20 breaths per minute or arterial carbon dioxide tension (PaCO2) of less than 32mm Hg, 4) abnormal white blood cell count (>12,000/µL or < 4,000/µL or >10% immature [band] forms). Septic shock was defined as sepsis associated with organ dysfunction and persistent hypotension despite volume replacement.

According to international guidelines, blood cultures were collected simultaneously from both central line and peripheral blood. So doing, five different mutually exclusive conditions were identified: 1) significant different time to positivization of blood cultures (at least 2 hours) between central line sample and peripheral sample (sepsis related to CVC - CLABSIs); 2) not significant different time to positivization of blood cultures (sepsis not related to CVC); 3) positive blood cultures from central line sample and negative from peripheral one (CVC colonization); 4) negative blood cultures from central line sample and positive from peripheral one (contaminated blood cultures); 5) negative blood cultures from both peripheral and central line samples (SIRS not sustained by sepsis). CVCs were removed when conditions 1 and 3 occurred. Catheter tips were collected and prepared for subsequent microbiological analysis and identified microbial species have been reported.

Each catheter was designated by type of vessel used (peripheral versus central); site of insertion (subclavian, femoral, internal jugular, peripheral, and Peripherally Inserted Central Catheter [PICC]).

Moreover, for each patient, data concerning provenance, parenteral nutrition, presence of tracheostomy tube and mechanical ventilation were collected.

Finally, in order to measure the severity of clinical condition of each patient, APACHE III score and Charlson's Comorbidity Index score were calculated.

Microbiological methods The entire medical center is served by a central microbiology laboratory, which is open from 7:00 AM to 7:00 PM, Monday through Saturday.

For adult patients with suspected BSIs, the center's standard of care requires the sequential collection at 30-min intervals of at least three sets of aerobic and anaerobic BCs (CLSI). For each set, a 20-mL blood sample is collected via a single venipuncture or intravascular line access. Skin or access ports are disinfected with alcohol and povidone iodine.

The blood sample is used to inoculate one BACTEC Plus Aerobic/F and Anaerobic bottles (10 mL of blood each) (Becton Dickinson Instrument Systems, Sparks, Md). The bottles are brought to the laboratory and incubated up to five days in the BACTEC FX automated blood culture instrument (Cultures arriving when the laboratory is closed are stored at room temperature in accordance with manufacturers' instructions). When the growth index of a bottle was positive, broth aliquots were collected for standard identification studies, which entailed Gram staining (the results of which were immediately reported to the patient's physician), routine subculture, and matrix-assisted laser desorption ionization-time of flight (MALDI-TOF) mass spectrometry (MALDI BioTyper, Bruker Daltonik GmbH, Leipzig, Germany) analysis of culture samples, supplemented when necessary with additional biochemical methods and/or 16S rRNA gene sequencing. Antibiotic susceptibility tests were performed using the Vitek 2 system (bioMérieux, Marcy l'Etoile, France). Confirmatory MIC testing for oxyimino-cephalosporins and carbapenems was carried out by Etest (bioMérieux). Results were interpreted according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) breakpoints (EUCAST table).

Study design The study was divided in two periods of equal duration time (9 months): a preliminary prospective observational period (phase I) and a subsequent prospective interventional period (phase II).

During phase II, two interventional strategies have been adopted:

1. at the beginning of interventional study and then every 45 days, physicians and nurses of RICU have been trained and retrained to GAVECELT ("Long Term Venous Central Lines" Open Group - www.gavecelt.it) "bundle" recommendations concerning the management of CVC. The bundle includes: hand hygiene and precautions for protection and safety, adequate insertion site, echo-guided placement of central venous line, use of clorexidine 2% for skin disinfection of insertion site chosen and subsequent continuous or discontinuous disinfection of exit site, use of suture-less devices, use of transparent semi-permeable dressing whenever applicable and immediate removal of catheter when no longer needed. Moreover, in order to reduce the use of unnecessary catheters, the investigators regularly evaluated the need for CVCs for both patients admitted to RICU and patients moved out of the ICU and unnecessary catheters were promptly removed.
2. After the first training meeting, the use of Curos® Disinfecting Port Protector for needleless valves port-protector (CUROS, 70% isopropyl alcohol-impregnated, Ivera Medical, San Diego, California, US) has been introduced.

Patients ruled in during the interventional period have been randomized into two groups:

1. patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations.
2. Patients with CVC managed by healthcare workers trained/retrained to GAVECELT recommendations with the aid of port protector devices.

Curos® Disinfecting Port Protector is a passive disinfection device that luer-locks securely onto needleless IV ports to disinfect in 3 minutes. If not removed, ports stay clean and protected for 7 days. The Curos® is intended for use on swabbable luer access valves as a disinfecting cleaner prior to line access and to act as a physical barrier to contamination between line accesses. Curos disinfects the valve three minutes after application and acts as a physical barrier to contamination for up to seven days if not removed.

ELIGIBILITY:
Inclusion Criteria:

* CVC placed during hospitalization in RICU;
* CVC already placed at admittance without signs of systemic inflammatory response syndrome (SIRS) during first 48h from admission to RICU;
* CVC already placed at admittance without evidence of microbiologic contamination of blood cultures;
* written informed consent.

Exclusion Criteria:

* CVC placed during hospitalization in other Hospital;
* CVC placed during hospitalization in other Unit with signs of systemic inflammatory response syndrome (SIRS) during first 48h from admission to RICU and / or evidence of microbiologic contamination of blood cultures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of CLABSIs. | Through study completion, an average of 18 months.
  Efficacy of educational interventions alone and combined with port protector as adjuvant tool on rate of CLABSIs.

SECONDARY OUTCOMES:
Rate of CVC colonizations | Through study completion, an average of 18 months.
  Efficacy of educational interventions alone and combined with port protector as adjuvant tool on rate of CVC colonizations.
Rate of contaminated blood cultures. | Through study completion, an average of 18 months.
  Efficacy of educational interventions alone and combined with port protector as adjuvant tool on rate of contaminated blood cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Inchingolo, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Gemelli, Catholic University of Sacred Heart; Giuseppe M Corbo, MD, Prof., Study Director — Fondazione Policlinico Universitario Gemelli, Catholic University of Sacred Heart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inchingolo R, Pasciuto G, Magnini D, Cavalletti M, Scoppettuolo G, Montemurro G, Smargiassi A, Torelli R, Sanguinetti M, Spanu T, Corbo GM, Richeldi L. Educational interventions alone and combined with port protector reduce the rate of central venous catheter infection and colonization in respiratory semi-intensive care unit. BMC Infect Dis. 2019 Mar 4;19(1):215. doi: 10.1186/s12879-019-3848-z. PMID 30832598